CLINICAL TRIAL: NCT01965730
Title: The Effect of Standard vs Aggressive Dosing Regimens for Epsilon-aminocaproic Acid on a Quantifiable Parameter of Fibrinolysis as Measured by Thromboelastography
Brief Title: Dosing of Amicar and Measure of Fibrinolysis by TEG During Cardiac Surgery
Acronym: EACA
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: the study was suspended due to shortage of the study drug (amicar).
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 816724
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Aortic Disease
Keywords: dilated ascending aorta
MeSH Terms: conditions — Aortic Diseases | interventions — Aminocaproic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- epsilon-aminocaproic acid (EACA) (Active Comparator): 75mg/kg loading dose with infusion 15mg/kg/hr
  Interventions: Drug: epsilon-aminocaproic acid (EACA)
- EACA (Experimental): 125mg/kg loading dose of EACA followed by an infusion of EACA at 25mg/kg/hr for length of cardiac surgery.
  Interventions: Drug: epsilon-aminocaproic acid (EACA)

INTERVENTIONS:
Drug: epsilon-aminocaproic acid (EACA)
  Other Names: Amicar

SUMMARY:
This study hopes to determine the optimal antifibrinolytic dosing to decrease bleeding and blood transfusion after cardiac surgery without increasing adverse events

ELIGIBILITY:
Inclusion Criteria:

* Ability to sign informed consent
* Elective cardiac surgery patients undergoing primary surgery involving circulatory arrest

Exclusion Criteria:

* Inability to sign informed consent
* Baseline hypercoagulable condition as defined in medical record
* Coronary disease with untreated lesions or recent coronary stent placement
* Severe renal dysfunction (ESRD) as documented in medical record

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
degree of fibrinolysis as measured by thromboelastography | Length of cardiac surgery
  The primary objective of the study will be to determine if a change in EACA dosing for cardiac surgery cases involving circulatory arrest actually leads to a quantifiable change in the degree of fibrinolysis as measured by TEG.

CONTACTS AND LOCATIONS:
Overall Officials: Prakash A Patel, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States